CLINICAL TRIAL: NCT06787066
Title: Sympathetic Vascular Transduction Across the Menopause Transition: Contributing Mechanisms
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Associate Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2125473
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Menopause
Keywords: Menopause; Sympathetic nerve activity; Sympathetic transduction; Blood flow; Women's health; Blood pressure
MeSH Terms: interventions — Propranolol; Phentolamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Women (Other): Women ages 18-70 years will participate.
  Interventions: Drug: Propranolol Hydrochloride; Drug: Phentolamine Injection

INTERVENTIONS:
Drug: Propranolol Hydrochloride — Examine how IV propranolol impacts sympathetic transduction
Drug: Phentolamine Injection — Examine how IV phentolamine impacts sympathetic transduction

SUMMARY:
The investigators aim to assess the interactions between the sympathetic nervous system and the vasculature in women across the menopause transition to better understand why aging women have a higher risk of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Assigned female at birth
* 18-70 years of age
* Body mass index (BMI) <30 kg/m2

Exclusion Criteria:

* Assigned male at birth
* Pregnancy, breastfeeding
* Body mass index ≥30 kg/m2
* Oral hormonal contraception in last 6 months, history of hormone replacement therapy, oophorectomy
* Current smoking/nicotine use
* Increased risk of bleeding, pro-coagulant disorders, clotting disorders, anticoagulation therapy
* Nerve/neurologic disease
* Cardiovascular, hepatic, renal, respiratory disease
* Blood pressure ≥140/90 mmHg
* Diabetes, Polycystic ovarian syndrome
* Communication barriers
* Prescription medications

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sympathetic transduction | 1 day (single study visit)
  Assessing the relative change in blood flow (Doppler ultrasound) following an increase in sympathetic nerve activity.

SECONDARY OUTCOMES:
Blood flow | 1 day (single study visit)
  Measuring femoral artery blood flow using Doppler ultrasound.
Muscle sympathetic nerve activity | 1 day (single study visit)
  Measuring the sympathetic nerve activity of the fibular nerve using a microelectrode .

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No